CLINICAL TRIAL: NCT04688060
Title: Assosiations Between Fear of Fall, Functional Ambulation Category and Quality of Life in Stroke Survivors
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Tugba Sahbaz, specialist doctor of physical medicine and rehabilitation, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: KAEK/2019.04.09
Record Dates: First submitted 2020-12-24; First posted 2020-12-29 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Fall
Keywords: fear of fall; quality of life; ambulation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- fallers: stroke duration of 6 months or more follow 3-step commands, were able to walk 10m with no physical assistance with or without any assistive device, and scoring ≥3 on Functional Ambulation Category, and physically able to complete the testing procedure Patients who have fallen 1 or more times since stroke
  Interventions: Diagnostic Test: Falls Efficacy Scale-International (FES-I)
- non-fallers: stroke duration of 6 months or more follow 3-step commands, were able to walk 10m with no physical assistance with or without any assistive device, and scoring ≥3 on Functional Ambulation Category, and physically able to complete the testing procedure.
  Patients who have not fallen 1 or more times since stroke
  Interventions: Diagnostic Test: Falls Efficacy Scale-International (FES-I)

INTERVENTIONS:
Diagnostic Test: Falls Efficacy Scale-International (FES-I) — The FES-1 was used to assess the fear of falling level of participants about falling during indoor or outdoor activities. It has 16 items scored on a four-point Likert scale. The Turkish validated version of the FES-I was used in this study. The total score (sum of the 16 responses) ranging from 16 to 64 points was used for data analysis. A higher score indicates better mobility performance. A cut-off score of 27 points on the 16- item FES-I was used to differentiate high concern for falling from low concern
  Other Names: Functional Ambulation Category (FAC); Stroke Impact Scale 3.0 (SIS)

SUMMARY:
Stroke is one of the most common causes of acquired adult disability. The stroke survivors have lots of mobility difficulties such as poor standing, decreased walking speed, balance disturbances, and increased risk of falls (1).

Falling is a major threat to stroke patients for physical injury. Fracture resulting from falling, could affect the rehabilitation potential and functional recovery (2,3).

After a stroke, falls are one of the most common medical complications with a 73% incidence within the six months (4). In addition to physical components, psychological factors related falling include fear of falling(5). Fear of falling is defined as persisting concern regarding falling and associated with many negative physical and psychological factors (6,7). It not only affects a simple health concern, but also avoidance of activities and a loss of confidence (8).

To determine the associating factors of fear of falling (FOF) and the correlations between FOF, functional ambulation category (FAC) and quality of life (QOL) on stroke patients.

DETAILED DESCRIPTION:
This study was a cross-sectional observational study. Each participant was assessed with standardized questionnaires and examined. Eighty six hemiplegic cronic stroke patients were recruited from our clinic from March 2018 to December 2020 with informed consent. We divided the participants into two groups; with fallers and non-fallers.

The inclusion criteria were stroke duration of 6 months or more follow 3-step commands, were able to walk 10m with no physical assistance with or without any assistive device, and scoring ≥3 on Functional Ambulation Category, and physically able to complete the testing procedure.

Exclusion criteria were other neurologic diagnosesor were medically unstable, lower-extremity fracture, or other surgical procedures during the last 6 months and were unable to provide consent.

All participants signed a written consent prior to participation in the study. The study was approved by the local institutional review board. The study was conducted in accordance with the Declaration of Helsinki ethical principles for human experimentation.

Demographic characteristics and medical history recorded by questionnaire included age, height, weight, comorbidities, number of medications, use of assistive device, date of stroke onset, and side of stroke, hemorrhagic or ischemic.

Falls history included number of falls during last 6 months or number of falls since the stroke onset, if stroke was less than 6 months prior. Fear of falling was assessed by asking subjects if they were afraid of falling (yes, no) and also ranking Falls Efficacy Scale-International (FES-I)(1).

Also functional ambulation levels, motor functions, spasticity and quality of life were assessed using Functional Ambulation Category (FAC), Brunnstrom staging, Modified Ashworth scale (MAS), Stroke Impact Scale 3.0 (SIS) (2-5).

1. Delbaere K, Close JC, Mikolaizak AS, Sachdev PS, Brodaty H, Lord SR. The Falls Efficacy Scale International (FES-I). A compre- hensive longitudinal validation study. Age Ageing 2010;39:210-216
2. Mehrholz J, Wagner K, Rutte K, Meissner D, Pohl M. Predictive validity and responsiveness of the functional ambulation category in hemiparetic patients after stroke. Arch Phys Med Rehabil 2007; 88:1314-1319
3. Hantal AÖ, Doğu B, Büyükavcı R, Kuran B. İnme etki ölçeği 3, 0: Türk toplumundaki inmeli hastalarda güvenilirlik ve geçerlilik çalışması. Türk Fiz Tıp Rehab Derg. 2014;60:106-16.
4. Ansari NN, Naghdi S, Younesian P, Shayeghan M, practice. Inter-and intrarater reliability of the Modified Modified Ashworth Scale in patients with knee extensor poststroke spasticity. Physiotherapy theory. 2008;24(3):205-13.
5. Brunnstrom S. Motor testing procedures in hemiplegia: based on sequential recovery stages. Physical therapy. 1966;46(4):357-75.

ELIGIBILITY:
Inclusion Criteria:

* stroke duration of 6 months or more
* follow 3-step commands
* were able to walk 10m with no physical assistance with or without any assistive device,
* scoring ≥3 on Functional Ambulation Category,
* physically able to complete the testing procedure.

Exclusion Criteria:

* other neurologic diagnosesor were medically unstable,
* lower-extremity fracture,
* other surgical procedures during the last 6 months
* were unable to provide consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: stroke duration of 6 months or more follow 3-step commands 18-65 years were able to walk 10m with no physical assistance with or without any assistive device
Sampling Method: Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-01-10 (Actual); Study Completion 2021-01-10 (Actual)

PRIMARY OUTCOMES:
Falls Efficacy Scale-International (FES-I) | basline
  assess the fear of falling level of participants about falling during indoor or outdoor activities minumum score 16 maximum score 64 low, moderate, and high concern (16-19, 20-27, and 28-64)

CONTACTS AND LOCATIONS:
Locations (1):
- Tuğba Şahbaz, Istanbul, Bakırköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Delbaere K, Close JC, Mikolaizak AS, Sachdev PS, Brodaty H, Lord SR. The Falls Efficacy Scale International (FES-I). A comprehensive longitudinal validation study. Age Ageing. 2010 Mar;39(2):210-6. doi: 10.1093/ageing/afp225. Epub 2010 Jan 8. PMID 20061508
- [Background] Mehrholz J, Wagner K, Rutte K, Meissner D, Pohl M. Predictive validity and responsiveness of the functional ambulation category in hemiparetic patients after stroke. Arch Phys Med Rehabil. 2007 Oct;88(10):1314-9. doi: 10.1016/j.apmr.2007.06.764. PMID 17908575
- [Background] Ansari NN, Naghdi S, Younesian P, Shayeghan M. Inter- and intrarater reliability of the Modified Modified Ashworth Scale in patients with knee extensor poststroke spasticity. Physiother Theory Pract. 2008 May-Jun;24(3):205-13. doi: 10.1080/09593980701523802. PMID 18569857
- [Background] Brunnstrom S. Motor testing procedures in hemiplegia: based on sequential recovery stages. Phys Ther. 1966 Apr;46(4):357-75. doi: 10.1093/ptj/46.4.357. No abstract available. PMID 5907254
- See also: Hantal AÖ, Doğu B, Büyükavcı R, Kuran B. İnme etki ölçeği 3, 0: Türk toplumundaki inmeli hastalarda güvenilirlik ve geçerlilik çalışması. Türk Fiz Tıp Rehab Derg. 2014;60:106-16. — http://www.ftrdergisi.com/uploads/sayilar/286/buyuk/106-116.pdf